CLINICAL TRIAL: NCT05216211
Title: The Effect of Caudal Block on Optic Nerve Sheath Diameter in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Optic nerve Caudal
Record Dates: First submitted 2021-12-09; First posted 2022-01-31 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Pain; Intracranial Hypertension
MeSH Terms: conditions — Pain, Postoperative; Intracranial Hypertension | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Caudal (Active Comparator): Caudal block with 1 ml / kg, % 0.25 bupivacaine
  Interventions: Drug: Bupivacaine Hydrochloride
- Group Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — 1 ml / kg, % 0.25 bupivacaine
  Arms: Group Caudal

SUMMARY:
Caudal epidural block has been a widely used regional anesthesia method, especially in pediatric surgery, to provide intraoperative and postoperative analgesia. Studies on non-invasive methods used for intracranial pressure measurement have shown that optic nerve sheath diameter is related to intracranial pressure. Optic nerve sheath diameter measurement has high diagnostic accuracy for detecting increased intracranial pressure in children. The aim of the study is to investigate the effect of the caudal block on optic nerve sheath diameter in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* circumcision,
* inguinal hernia,
* undescended testis,
* hydrocele operation

Exclusion Criteria:

* neurological or spinal anomaly,
* coagulopathy
* allergy to local anesthetics,
* local infection in the area to be intervention,
* with increased intracranial pressure
* children with any ophthalmic pathology

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Optic Nerve Diameter | First minute
  Consecutive Optic Nerve Sheath Diameter Measurement from Both Eyes
Optic Nerve Diameter | 5th minutes
  Consecutive Optic Nerve Sheath Diameter Measurement from Both Eyes
Optic Nerve Diameter | 15th minutes
  Consecutive Optic Nerve Sheath Diameter Measurement from Both Eyes
Optic Nerve Diameter | 30th minutes
  Consecutive Optic Nerve Sheath Diameter Measurement from Both Eyes

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University School of Medicine, Erzurum, Yakutiye, Turkey (Türkiye)